CLINICAL TRIAL: NCT01259570
Title: Bioavailability of Vitamin D Encapsulated in Casein Micelles, Compared to Its Bioavailability in the Milk-fat, or in a Synthetic Emulsifier Currently Used for Supplementation and Enrichment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sophia Ish-Shalom, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3000007066
Record Dates: First submitted 2010-12-12; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Skimmilk enriched with VD encapsulated in CM (Active Comparator)
  Interventions: Dietary Supplement: Group 1
- VD will be dissolved in milkfat and homogenized into skimmilk (Active Comparator): VD will be dissolved in milkfat and homogenized into skimmilk
  Interventions: Dietary Supplement: Group 2
- 3% fat milk wherein the VD will be in CM (Active Comparator): 3% fat milk wherein the VD will be in CM
  Interventions: Dietary Supplement: group 3
- Placebo: un-enriched skimmilk. (Active Comparator): Placebo: un-enriched skimmilk.
  Interventions: Dietary Supplement: Group 4

INTERVENTIONS:
Dietary Supplement: Group 1 — Skimmilk enriched with VD encapsulated in CM
  Arms: Skimmilk enriched with VD encapsulated in CM
Dietary Supplement: Group 2 — VD will be dissolved in milkfat and homogenized into skimmilk
  Arms: VD will be dissolved in milkfat and homogenized into skimmilk
Dietary Supplement: group 3 — 3% fat milk wherein the VD will be in CM
  Arms: 3% fat milk wherein the VD will be in CM
Dietary Supplement: Group 4 — Placebo: un-enriched skimmilk.
  Arms: Placebo: un-enriched skimmilk.

SUMMARY:
The encapsulation within CM may improve bioavailability (BA) of vitamin D (VD), even in absence of fat.

As a model the investigators have chosen nonfat yoghurt. The investigators will prepare yoghurts from 4 milks: (1) Skimmilk enriched with 50,000 IU/150gr VD encapsulated in CM2 ; (2) 3% fat milk wherein same dose of VD - dissolved in milk fat and homogenized into skimmilk; (3) 3% fat milk wherein VD, at same dose, will be in CM; (4) Placebo: unenriched skimmilk. 120 healthy adults aged 18-65 will randomized to 5 groups and receive 150 gr yoghurt. Blood will be drawn before ingestion and on days 1,7,14. 25(OH)D will be det. by CMIA. In vitro simulated digestion will be studied.

Expected results: The BA of VD in CM would not be lower than in fat

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Metabolic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Bioavailability of vitamin D encapsulated in casein micelles, compared to its bioavailability in the milk-fat. | 1 year
  As a model we have chosen nonfat yoghurt. We will prepare yoghurts from 4 milks: (1) Skimmilk enriched with 50,000 IU/150gr VD encapsulated in CM2 ; (2) 3% fat milk wherein same dose of VD - dissolved in milk fat and homogenized into skimmilk; (3) 3% fat milk wherein VD, at same dose, will be in CM; (4) Placebo: unenriched skimmilk. 120 healthy adults aged 18-65 will randomized to 5 groups and receive 150 gr yoghurt. Blood will be drawn before ingestion and on days 1,7,14. 25(OH)D will be det. by